CLINICAL TRIAL: NCT03567057
Title: A Multicenter, Open-Label Safety and Efficacy Study of ADS-5102 Amantadine Extended Release Capsules in Patients With Multiple Sclerosis and Walking Impairment
Brief Title: A Safety and Efficacy Study of ADS-5102 in Patients With Multiple Sclerosis and Walking Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adamas Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADS-AMT-MS303
Record Dates: First submitted 2018-05-22; First posted 2018-06-25 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis; Walking Impairment
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADS-5102, 274 mg (Experimental): 274 mg ADS-5102, administered once daily at bedtime for up to 52 weeks
  Interventions: Drug: ADS-5102, 274 mg

INTERVENTIONS:
Drug: ADS-5102, 274 mg — Oral capsules
  Other Names: amantadine extended release

SUMMARY:
This study assessed the long-term safety and tolerability of ADS-5102 in subjects with MS and walking impairment who had completed the double-blind, placebo-controlled study of ADS-5102 in subjects with MS (ADS-AMT-301).

DETAILED DESCRIPTION:
This was a multicenter, open-label study of ADS-5102 (amantadine) extended-release capsules in subjects with MS and walking impairment who completed study drug treatment for 16 weeks and completed a Week 16 visit in Study ADS-AMT-MS301.

All enrolled subjects were to receive ADS-5102 at 137 mg for the first week, 205.5 mg for the second week, and 274 mg for the remainder of the 52-week open-label treatment period.

Subjects returned to the clinic for safety and efficacy assessments at Weeks 4, 24, and 52. In addition, a telephone visit for safety assessments was conducted at Week 2 and Week 38. Subjects who withdrew from the study prior to completion of the Week 52 visit had an early termination (ET) visit that included safety and efficacy assessments. Subjects who completed 52 weeks of open-label treatment had a final visit for post-treatment safety follow-up and efficacy assessment at Week 54.

All study visits and efficacy assessments were to be scheduled to occur at approximately the same time of day for each individual subject. Each subject's efficacy assessment was to be performed by the same clinical rater, if possible.

ELIGIBILITY:
Inclusion Criteria:

* Signed a current IRB-approved informed consent form
* Successful completion of a prior double blind study of ADS-5102 in patients with MS walking impairment.

Exclusion Criteria:

* Based on the judgment of the investigator or Medical Monitor, participation in the study would jeopardize the safety of the subject.
* If female, is pregnant or lactating
* If a sexually active female, is not surgically sterile or at least 2 years post-menopausal, or does not agree to utilize a highly effective hormonal method of contraception (an IUD, or vasectomized male partner is also acceptable), in combination with a barrier method, from baseline through at least 4 weeks after the completion of study treatment. If a sexually active male, does not agree to utilize condoms from screening through at least 4 weeks after the completion of study treatment.
* Anticipated treatment with any amantadine formulation other than ADS-5102
* Planned participation in another interventional clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2021-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Chief Medical Officer, MD, Study Director — Adamas Pharmaceuticals, Inc.
Locations (88):
- United States (78):
  - Adamas Clinical Site, Cullman, Alabama
  - Adamas Clinical Site, Phoenix, Arizona
  - Adamas Clinical Site, Tucson, Arizona
  - Adamas Clinical Site, Carlsbad, California
  - Adamas Clinical Site, Fresno, California
  - Adamas Clinical Site, Fullerton, California
  - Adamas Clinical Site, Long Beach, California
  - Adamas Clinical Site, Newport Beach, California
  - Adamas Clinical Site, Sacramento, California
  - Adamas Clinical Site, Aurora, Colorado
  - Adamas Clinical Site, Colorado Springs, Colorado
  - Adamas Clinical Site, Denver, Colorado
  - Adamas Clinical Site, Fort Collins, Colorado
  - Adamas Clinical Site, Fairfield, Connecticut
  - Adamas Clinical Site, New London, Connecticut
  - Adamas Clinical Site, Washington D.C., District of Columbia
  - Adamas Clinical Site, Maitland, Florida
  - Adamas Clinical Site, Miami, Florida
  - Adamas Clinical Site, Naples, Florida
  - Adamas Clinical Site, Orlando, Florida
  - Adamas Clinical Site, Ormond Beach, Florida
  - Adamas Clinical Site, Palm Coast, Florida
  - Adamas Clinical Site, Port Charlotte, Florida
  - Adamas Clinical Site, Sarasota, Florida
  - Adamas Clinical Site, St. Petersburg, Florida
  - Adamas Clinical Site, Tampa, Florida
  - Adamas Clinical Site, Vero Beach, Florida
  - Adamas Clinical Site, Atlanta, Georgia
  - Adamas Clinical Site, Savannah, Georgia
  - Adamas Clinical Site, Northbrook, Illinois
  - Adamas Clinical Site, Indianapolis, Indiana
  - Adamas Clinical Site, Kansas City, Kansas
  - Adamas Clinical Site, Lenexa, Kansas
  - Adamas Clinical Site, Overland Park, Kansas
  - Adamas Clinical Site, Burlington, Massachusetts
  - Adamas Clinical Site, Foxborough, Massachusetts
  - Adamas Clinical Site, Worcester, Massachusetts
  - Adamas Clinical Site, Detroit, Michigan
  - Adamas Clinical Site, Farmington Hills, Michigan
  - Adamas Clinical Site, Golden Valley, Minnesota
  - Adamas Clinical Site, Kansas City, Missouri
  - Adamas Clinical Site, St Louis, Missouri
  - Adamas Clinical Site, Great Falls, Montana
  - Adamas Clinical Site, Lincoln, Nebraska
  - Adamas Clinical Site, Omaha, Nebraska
  - Adamas Clinical Site, Las Vegas, Nevada
  - Adamas Clinical Site, Albuquerque, New Mexico
  - Adamas Clinical Site, Amherst, New York
  - Adamas Clinical Site, Lake Success, New York
  - Adamas Clinical Site, New York, New York
  - Adamas Clinical Site, Patchogue, New York
  - Adamas Clinical Site, Plainview, New York
  - Adamas Clinical Site, Rochester, New York
  - Adamas Clinical Site, Staten Island, New York
  - Adamas Clinical Site, Charlotte, North Carolina
  - Adamas Clinical Site, Raleigh, North Carolina
  - Adamas Clinical Site, Centerville, Ohio
  - Adamas Clinical Site, Cleveland, Ohio
  - Adamas Clinical Site, Columbus, Ohio
  - Adamas Clinical Site, Oklahoma City, Oklahoma
  - Adamas Clinical Site, Portland, Oregon
  - Adamas Clinical Site, Philadelphia, Pennsylvania
  - Adamas Clinical Site, Charleston, South Carolina
  - Adamas Clinical Site, Greer, South Carolina
  - Adamas Clinical Site, Rock Hill, South Carolina
  - Adamas Clinical Site, Spartanburg, South Carolina
  - Adamas Clinical Site, Cordova, Tennessee
  - Adamas Clinical Site, Franklin, Tennessee
  - Adamas Clinical Site, Johnson City, Tennessee
  - Adamas Clinical Site, Houston, Texas
  - Adamas Clinical Site, Lubbock, Texas
  - Adamas Clinical Site, Round Rock, Texas
  - Adamas Clinical Site, Salt Lake City, Utah
  - Adamas Clinical Site, Newport News, Virginia
  - Adamas Clinical Site, Norfolk, Virginia
  - Adamas Clinical Site, Kirkland, Washington
  - Adamas Clinical Site, Seattle, Washington
  - Adamas Clinical Site, Milwaukee, Wisconsin
- Canada (10):
  - Adamas Clinical Site, Edmonton, Alberta
  - Adamas Clinical Site, Lethbridge, Alberta
  - Adamas Clinical Site, Burnaby, Brithis Columbia
  - Adamas Clinical Site, Vancouver, British Columbia
  - Adamas Clinical Site, Hamilton, Ontario
  - Adamas Clinical Site, London, Ontario
  - Adamas Clinical Site, Ottawa, Ontario
  - Adamas Clinical Site, Greenfield Park, Quebec
  - Adamas Clinical Site, Montreal, Quebec
  - Adamas Clinical Site, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/274 mg ADS-5102: Consists of subjects who received placebo in Study ADS-AMT-MS301 and 274 mg ADS-5102 in the current study (ADS-AMT-MS303)
- 137 mg ADS-5102/274 mg ADS-5102: Consists of subjects who received 137 mg ADS-5102 in Study ADS-AMT-MS301 and 274 mg ADS-5102 in the current study (ADS-AMT-MS303)
- 274 mg ADS-5102/274 mg ADS-5102: Consists of subjects who 274 mg ADS-5102 in both Studies ADS-AMT-MS301 and ADS-AMT-MS303
Period: Overall Study
Arm/Group | Placebo/274 mg ADS-5102 | 137 mg ADS-5102/274 mg ADS-5102 | 274 mg ADS-5102/274 mg ADS-5102
Started | 159 | 151 | 114
Completed | 64 | 64 | 68
Not Completed | 95 | 87 | 46
Not completed — Adverse Event | 56 | 53 | 28
Not completed — Withdrawal by Subject | 22 | 24 | 13
Not completed — Lost to Follow-up | 3 | 5 | 2
Not completed — COVID-19 pandemic | 4 | 3 | 0
Not completed — Non-compliance with study drug | 4 | 2 | 0
Not completed — Lack of Efficacy | 3 | 0 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Unstable medical condition | 1 | 0 | 0
Not completed — Medical history event | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/274 mg ADS-5102 | 137 mg ADS-5102/274 mg ADS-5102 | 274 mg ADS-5102/274 mg ADS-5102 | Total
Number analyzed (Participants) | 159 | 151 | 114 | 424
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (9.80) | 54.8 (9.12) | 53.0 (9.40) | 54.3 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 100 | 76 | 284
  Male | 51 | 51 | 38 | 140
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 20 | 20 | 12 | 52
  White | 133 | 128 | 99 | 360
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 2 | 2 | 3 | 7
Baseline T25FW [Count of Participants; unit: Participants]
  <Median of enrolled population (9.4 seconds) | 63 | 85 | 58 | 206
  >Median of enrolled population (9.4 seconds) | 96 | 66 | 55 | 217
  Missing | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events
Description: The incidence of treatment-emergent adverse events was used as the measure for long-term safety and tolerability of ADS-5102.
Time Frame: Through study completion, an average of 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/274 mg ADS-5102 | 137 mg ADS-5102/274 mg ADS-5102 | 274 mg ADS-5102/274 mg ADS-5102
Number analyzed (Participants) | 159 | 151 | 114
Participants | 122 | 116 | 86

2. Secondary Outcome: Timed 25-Foot Walk (Feet/Second) (Baseline Value)
Description: The timed 25-foot walk is a measure of lower extremity function. The subject is directed to a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The task is immediately administered again by having the subject walk back the same distance. The result is reported as speed (feet per second). Improvement is indicated by an increase in speed.
Time Frame: Baseline
Population: Modified intent-to-treat: subjects with available data
Measure: Mean (Standard Deviation); unit: feet/second
Arm/Group | Placebo/274 mg ADS-5102 | 137 mg ADS-5102/274 mg ADS-5102 | 274 mg ADS-5102/274 mg ADS-5102
Number analyzed (Participants) | 159 | 151 | 113
feet/second | 2.43 (0.853) | 2.68 (0.840) | 2.66 (0.878)

3. Secondary Outcome: Timed 25-Foot Walk (Feet/Second) (Week 24 Value)
Description: as for outcome 2
Time Frame: 24 weeks
Population: Modified intent-to-treat: subjects with available data
Measure: Mean (Standard Deviation); unit: feet/second
Arm/Group | Placebo/274 mg ADS-5102 | 137 mg ADS-5102/274 mg ADS-5102 | 274 mg ADS-5102/274 mg ADS-5102
Number analyzed (Participants) | 84 | 89 | 74
feet/second | 2.50 (0.832) | 2.72 (0.969) | 2.71 (0.957)

4. Secondary Outcome: Timed 25-Foot Walk (Feet/Second) (Week 52 Value)
Description: as for outcome 2
Time Frame: 52 weeks
Population: Modified intent-to-treat: subjects with available data
Measure: Mean (Standard Deviation); unit: feet/second
Arm/Group | Placebo/274 mg ADS-5102 | 137 mg ADS-5102/274 mg ADS-5102 | 274 mg ADS-5102/274 mg ADS-5102
Number analyzed (Participants) | 58 | 57 | 59
feet/second | 2.35 (0.900) | 2.68 (1.055) | 2.65 (0.996)

5. Secondary Outcome: Timed up and go (Baseline Value)
Description: The "timed up and go" is a measure of lower extremity strength, balance, and coordination. The subject stands up from a chair, walks 3 meters then turns around and walks back to the chair to sit down. The result is reported in seconds. Improvement is indicated by negative change scores.
Time Frame: Baseline
Population: Modified intent-to-treat population: subjects with available data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo/274 mg ADS-5102 | 137 mg ADS-5102/274 mg ADS-5102 | 274 mg ADS-5102/274 mg ADS-5102
Number analyzed (Participants) | 159 | 151 | 113
seconds | 17.60 (8.516) | 16.89 (17.536) | 16.80 (10.652)

6. Secondary Outcome: Timed up and go (Week 24 Value)
Description: as for outcome 5
Time Frame: 24 weeks
Population: Modified intent-to-treat population: subjects with available data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo/274 mg ADS-5102 | 137 mg ADS-5102/274 mg ADS-5102 | 274 mg ADS-5102/274 mg ADS-5102
Number analyzed (Participants) | 84 | 88 | 74
seconds | 17.39 (9.466) | 15.36 (9.109) | 16.89 (11.649)

7. Secondary Outcome: Timed up and go (Week 52 Value)
Description: as for outcome 5
Time Frame: 52 weeks
Population: Modified intent-to-treat population: subjects with available data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo/274 mg ADS-5102 | 137 mg ADS-5102/274 mg ADS-5102 | 274 mg ADS-5102/274 mg ADS-5102
Number analyzed (Participants) | 57 | 57 | 59
seconds | 18.68 (11.710) | 15.92 (11.820) | 17.37 (12.311)

8. Secondary Outcome: 2-Minute Walk Test (Baseline Value)
Description: The 2-Minute Walk test is a measure of lower extremity function. The subject is instructed to walk as far as possible in 2 minutes, and the distance is measured in meters. Improvement is indicated by positive change scores.
Time Frame: Baseline
Population: Modified intent-to-treat: subjects with available data
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo/274 mg ADS-5102 | 137 mg ADS-5102/274 mg ADS-5102 | 274 mg ADS-5102/274 mg ADS-5102
Number analyzed (Participants) | 159 | 150 | 112
meters | 80.26 (31.899) | 89.99 (31.679) | 87.31 (31.351)

9. Secondary Outcome: 2-Minute Walk Test (Week 24 Value)
Description: as for outcome 8
Time Frame: 24 weeks
Population: Modified intent-to-treat: subjects with available data
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo/274 mg ADS-5102 | 137 mg ADS-5102/274 mg ADS-5102 | 274 mg ADS-5102/274 mg ADS-5102
Number analyzed (Participants) | 83 | 87 | 71
meters | 81.48 (31.653) | 87.99 (34.195) | 92.03 (38.371)

10. Secondary Outcome: 2-Minute Walk Test (Week 52 Value)
Description: as for outcome 8
Time Frame: 52 weeks
Population: Modified intent-to-treat: subjects with available data
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo/274 mg ADS-5102 | 137 mg ADS-5102/274 mg ADS-5102 | 274 mg ADS-5102/274 mg ADS-5102
Number analyzed (Participants) | 58 | 55 | 57
meters | 77.45 (34.147) | 89.18 (36.707) | 89.14 (37.295)

ADVERSE EVENTS:
Time Frame: Approximately 1 year.
Arm/Group | Placebo/274 mg ADS-5102 | 137 mg ADS-5102/274 mg ADS-5102 | 274 mg ADS-5102/274 mg ADS-5102
All-Cause Mortality (participants affected / at risk) | 1/159 | 0/151 | 0/114
Serious Adverse Events (participants affected / at risk) | 20/159 | 20/151 | 7/114
Other Adverse Events (participants affected / at risk) | 122/159 | 116/151 | 86/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/274 mg ADS-5102 (N=159) | 137 mg ADS-5102/274 mg ADS-5102 (N=151) | 274 mg ADS-5102/274 mg ADS-5102 (N=114)
Multiple sclerosis relapse (Nervous system disorders) | 3 | 2 | 0
Encephalopathy (Nervous system disorders) | 1 | 1 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1
Uhthoff's phenomenon (Nervous system disorders) | 1 | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Generalized tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Sepsis (Infections and infestations) | 1 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1
Bursitis infective staphylococcal (Infections and infestations) | 0 | 0 | 1
Pharyngeal abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Viral sepsis (Infections and infestations) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Catatonia (Psychiatric disorders) | 0 | 1 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/274 mg ADS-5102 (N=159) | 137 mg ADS-5102/274 mg ADS-5102 (N=151) | 274 mg ADS-5102/274 mg ADS-5102 (N=114)
Multiple sclerosis relapse (Nervous system disorders) | 11 | 8 | 8
Dizziness (Nervous system disorders) | 8 | 8 | 3
Headache (Nervous system disorders) | 5 | 7 | 6
Balance disorder (Nervous system disorders) | 8 | 2 | 1
Oedema peripheral (General disorders) | 28 | 17 | 10
Peripheral swelling (General disorders) | 9 | 4 | 2
Urinary tract infection (Infections and infestations) | 16 | 15 | 15
Hallucination, visual (Psychiatric disorders) | 7 | 11 | 4
Insomnia (Psychiatric disorders) | 5 | 10 | 5
Dry mouth (Gastrointestinal disorders) | 13 | 18 | 2
Constipation (Gastrointestinal disorders) | 15 | 9 | 5
Livedo reticularis (Skin and subcutaneous tissue disorders) | 10 | 18 | 8
Fall (Injury, poisoning and procedural complications) | 14 | 16 | 17
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT03567057/Prot_SAP_000.pdf